# STATISTICAL ANALYSIS PLAN PHASE 2

# FINAL DATE OF PLAN:

14Dec2016

# **STUDY DRUG:**

NBI-98854

# **PROTOCOL NUMBER:**

NBI-98854-1505

# **STUDY TITLE:**

A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of NBI-98854 in Adult Subjects with Tourette Syndrome

# **SPONSOR:**

Neurocrine Biosciences, Inc. 12780 El Camino Real San Diego, CA 92130

Telephone: (858) 617-7600

**CONFIDENTIAL** 

# SIGNATURE PAGE

# TABLE OF CONTENTS

| LIST OF | ABBREVIATIONS | 6 |
|---|---|---|
| 1. | INTRODUCTION | 8 |
| 2. | STUDY OBJECTIVES | 8 |
| 2.1. | Study Design and Assessments | 8 |
| 3. | STATISTICAL ANALYSES | 10 |
| 3.1. | General Statistical Procedures | 10 |
| 3.2. | Sample Size Calculation | 10 |
| 3.3. | Pooling of Sites | 11 |
| 3.4. | Handling of Early Termination Visit Data | 11 |
| 3.5. | Handling of Missing Data. | 11 |
| 3.5.1. | Missing and incomplete dates | 12 |
| 3.6. | Coding Dictionary | 12 |
| 3.7. | Analysis Sets | 13 |
| 3.7.1. | Definition of Analysis Sets | 13 |
| 3.7.2. | Summary of Analysis Sets | 13 |
| 3.7.3. | Application of Analysis Sets | 13 |
| 3.8. | Subject Randomization and Disposition | 14 |
| 3.9. | Important Protocol Deviations. | 14 |
| 3.10. | Demographic Data and Baseline Characteristics | 15 |
| 3.11. | Medical History | 15 |
| 3.12. | Study Drug Dosing Compliance | 15 |
| 3.13. | Dose Reduction Summary | 16 |
| 3.14. | Pharmacokinetic Data | 16 |
| 3.15. | Efficacy Data | 17 |
| 3.15.1. | Efficacy Endpoints | 17 |
| 3.15.2. | Primary Efficacy Endpoint | 18 |
| 3.15.3. | Key Secondary Efficacy Endpoint | 20 |
| 3.15.4. | Fixed-Sequence Testing Procedure to Control for Multiple Comparisons | 20 |
| 3.15.5. | Sensitivity Analyses for Primary Efficacy Endpoint | 21 |
| 3.15.6. | Secondary Efficacy Endpoints | 23 |
| 3 15 6 1 | VGTSS TTS Responder Analysis | 23 |

# Neurocrine Biosciences, Inc.

# NBI-98854-1505 Statistical Analysis Plan

| 3.15.6.2. | YGTSS Impairment Score | 24 |
|---|---|---|
| 3.15.6.3. | YGTSS Global Tic Severity Score | 24 |
| 3.15.6.4. | Rush Video-based Tic Rating Scale (RTRS) | 25 |
| 3.15.6.5. | Premonitory Urge for Tics Scale (PUTS) | 25 |
| 3.15.6.6. | CGI-Tics-Severity | 26 |
| 3.15.6.7. | CGI-TS-Improvement Responder Analysis | 27 |
| 3.16. | Safety Data | 27 |
| 3.16.1. | Adverse Events | 27 |
| 3.16.1.1. | Adverse Event Overall Summary | 28 |
| 3.16.1.2. | Adverse Events Resulting in Study Drug Dose Reductions | 28 |
| 3.16.1.3. | Adverse Events Resulting in Premature Study Discontinuation | 28 |
| 3.16.1.4. | Deaths and Other Serious Adverse Events | 28 |
| 3.16.2. | Clinical Laboratory Data | 29 |
| 3.16.3. | Physical Examination and Weight | 31 |
| 3.16.4. | Vital Signs | 31 |
| 3.16.5. | Electrocardiogram | 31 |
| 3.16.6. | Columbia-Suicide Severity Rating Scale (C-SSRS) | 32 |
| 3.16.7. | Extrapyramidal Symptom Rating Scale-Abbreviated (ESRS-A) | 33 |
| 3.16.8. | Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 34 |
| 3.16.9. | Structured Interview Guide for the Hamilton Depression Rating Scale (SIGH-D-17) | 34 |
| 3.16.10. | Prior and Concomitant Medications | 35 |
| 3.17. | Additional Data Presentations | 35 |
| 3.17.1. | Inclusion and Exclusion Criteria | 35 |
| 3.17.2. | Serology Test Results | 35 |
| 3.17.3. | Pregnancy Test Results. | 35 |
| 3.17.4. | Urine Drug Screen and Alcohol Breath Test | 36 |
| 4. | DEVIATIONS FROM PROTOCOL PLANNED ANALYSIS | 36 |
| 5. | PERFORMANCE QUALIFICATION OF SAS® PROGRAMS | 36 |
| 6. | REFERENCES | 37 |

# LIST OF TABLES

| Table 1: | Allowable Study Day Range for Early Termination Visit Mapping | 11 |
|---|---|---|
| Table 2: | Data Summaries by Analysis Set. | 14 |
| Table 3: | Efficacy Endpoints and Classification | 18 |
| Table 4: | Potential Clinically Significant Criteria for Clinical Laboratory Variables | 30 |
| Table 5: | Potentially Clinically Significant Criteria for Vital Signs | 31 |

### LIST OF ABBREVIATIONS

Abbreviation **Term** AΕ Adverse event ALT Alanine aminotransferase ANCOVA Analysis of covariance ANOVA Analysis of variance AST Aspartate aminotransferase ATC Anatomical Therapeutic Chemical Classification BLQ Below the limit of quantification **BOCF** Baseline observation carried forward Clinical Global Impression of Tics **CGI-Tics** CGI-TS Clinical Global Impression of Change – Tourette Syndrome Columbia-Suicide Severity Rating Scale C-SSRS CYP2D6 Cytochrome P450 2D6 **ECG** Electrocardiogram eCRF Electronic case report form Extrapyramidal Symptom Rating Scale - Abbreviated **ESRS-A** ET Early termination GGT Gamma-glutamyl transferase HBsAg Hepatitis B surface antigen **HCV-Ab** Hepatitis C antibody HIV-Ab Human immunodeficiency virus antibody **IPD** Important protocol deviation ITT Intent-to-treat J2R Jump to reference LS Least squares MAR Missing at random MedDRA Medical Dictionary for Regulatory Activities MMRM Mixed-effect model repeated measures n, N Sample size (number of subjects) Neurocrine Biosciences, Inc. NBI **PCS** Potentially Clinically Significant PK Pharmacokinetic(s) PP Per-protocol

| Abbreviation | Term |
|---|---|
| PT | Preferred term |
| PUTS | Premonitory Urge for Tics Scale |
| QTcF | Fridericia's correction of QT interval |
| RTRS | Rush Video-Based Tic Rating Scale |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| $\mathrm{SAS}^{\circledR}$ | SAS® statistical software |
| SD | Standard deviation |
| SEM | Standard error of the mean |
| SIGH-D-17 | Structured Interview Guide for the Hamilton Depression Rating Scale, 17-Item |
| SOC | System organ class |
| TEAE | Treatment-emergent adverse event |
| TS | Tourette Syndrome |
| TTS | Total Tic Score |
| WHO | World Health Organization |
| Y-BOCS | Yale-Brown Obsessive-Compulsive Scale |
| YGTSS | Yale Global Tic Severity Scale |

### 1. INTRODUCTION

This statistical analysis plan (SAP) provides a detailed description of the analyses, tables, figures, and listings that will be prepared to summarize the data from the Phase 2 study described in Neurocrine Biosciences, Inc. (NBI) Protocol NBI-98854-1505.

### 2. STUDY OBJECTIVES

The objectives of this clinical study are as follows:

- To evaluate the efficacy of 2 active doses of NBI-98854 (40 mg and 80 mg) administered once daily in adult subjects with Tourette syndrome (TS).
- To assess the safety and tolerability of repeated daily doses of NBI-98854 in adult subjects with TS.
- To evaluate plasma exposure of NBI-98854 and its metabolite, NBI-98782, following repeated daily doses of NBI-98854.

# 2.1. Study Design and Assessments

This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel group study in a total of approximately 90 male and female subjects, 18 to 64 years of age, with a Diagnostic and Statistical Manual of Mental Disorders, 4th or 5th Editions, diagnosis of TS.

After providing informed consent, subjects will be screened to determine eligibility within 21 days (Days -21 to -1) before the start of study drug dosing on Day 1. Subjects may also be asked to sign an optional release form to allow their Rush Video-based Tic Rating Scale (RTRS) video recordings to be used for educational purposes.

On Day -1 (baseline), eligible subjects will return to the study center for collection of baseline safety and efficacy assessments and collection of a blood sample for subsequent determination of their cytochrome P450 2D6 (CYP2D6) metabolizer status. Subjects who continue to be eligible for the study will then be randomized (1:1:1) to placebo or 1 of 2 active doses of NBI-98854 (40 mg or 80 mg). A 2-week supply of study drug will be dispensed. Study drug will be administered in a double-dummy fashion throughout the 8-week double-blind treatment period. Beginning on Day 1, study drug will be administered at home once daily in the morning with a standard breakfast through Week 8. The NBI-98854 80 mg dose will be titrated in a blinded fashion (subjects will receive 40 mg for the first week followed by 80 mg).

At any time, if the subject is unable to tolerate their current dose, the investigator may decrease the subject's dose. The investigator is allowed to reduce the subject's dose only one time during the study. Subjects who have had a dose reduction and are unable to tolerate the new dose will be discontinued from the study. To maintain the study blind, subjects receiving 40 mg or placebo who have a dose reduction will continue to receive their current dose and subjects receiving 80 mg will be reduced to 40 mg.

During the double-blind treatment period, subjects will return to the study center at 2-week intervals (end of Weeks 2, 4, 6, and 8) for study assessments and dispensing of study drug

(Weeks 2, 4, and 6 only). All subjects who have completed the 8-week treatment period will enter a 2-week follow-up period with a follow-up visit at Week 10 (or early termination).

Efficacy assessments for TS symptomatology include the Total Tic Score (TTS) from the Yale Global Tic Severity Scale (YGTSS) as the primary efficacy variable, and the YGTSS Impairment and Global Tic Severity scores, the Rush Video-Based Tic Rating Scale (RTRS), the Premonitory Urge for Tics Scale (PUTS), the Clinical Global Impression of Change-Tourette Syndrome (CGI-TS)-Improvement scale, and the Clinical Global Impression of Tics (CGI-Tics)-Severity scale as secondary efficacy variables. The YGTSS, RTRS, and PUTS will be administered at screening, on Day -1 (the day before dosing), during the double-blind treatment period (Weeks 2, 4, 6, and 8), and at the follow-up visit (Week 10) or early termination. Note that all efficacy analyses for YGTSS-related variables are based on the certified site rater scores. Computer-generated tandem scores are also collected in the study database and will be presented in data listings only.

The CGI-Tics-Severity will be evaluated at screening and Day -1 (baseline), and then both the CGI-Tics-Severity and CGI-TS-Improvement scales will be administered at Weeks 2, 4, 6, and 8 and at the follow-up visit (Week 10) or early termination.

Safety assessments will also be collected at scheduled times throughout the study, including adverse event (AE) monitoring, clinical laboratory tests (hematology, clinical chemistry, and urinalysis), vital sign measurements, physical examinations (including weight), electrocardiograms (ECGs), Columbia Suicide Severity Rating Scale (C-SSRS), Extrapyramidal Symptom Rating Scale-Abbreviated (ESRS-A; note that this assessment was added in study protocol amendment 3 and therefore, is not available for all subjects at all visits), Structured Interview Guide for the Hamilton Depression Rating Scale, 17-Item (SIGH-D-17), and the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS).

Blood samples for plasma drug concentration and metabolite analyses will be collected during the treatment period (end of Weeks 2, 4, 6, and 8), and at the follow-up visit (Week 10) or early termination).

### 3. STATISTICAL ANALYSES

All analyses described in this plan are considered *a priori* analyses in that they have been defined prior to locking the study database. Analyses defined subsequent to locking the database will be considered *post hoc* analyses and will be applied as exploratory methodology. Any *post hoc* analyses will be clearly identified in the clinical study report.

### 3.1. General Statistical Procedures

Descriptive and inferential statistical methods will be used to summarize the data from this study. The term "descriptive statistics" refers to the number of subjects (n), mean, median, standard deviation (SD), standard error of the mean (SEM), minimum, and maximum for continuous variables; and refers to the number and/or percentage of subjects (or events) for categorical variables. The term "inferential statistics" refers to hypothesis tests which will be performed to assess differences between each NBI-98854 treatment (dose) group and the placebo group for selected efficacy variables. All hypothesis tests will be tests of the null hypothesis of no difference between the treatment groups being compared versus the two-sided alternative hypothesis that there is a difference.

The primary efficacy endpoint in this study is the YGTSS TTS mean change from baseline (Day -1) to Week 8 based on the certified site rater scores. Inferential statistics will be calculated for this endpoint as well as for secondary and exploratory efficacy endpoints. Two-sided p-values will be reported for all hypothesis tests; however, interpretation of the p-values for the primary and key secondary efficacy endpoints will be based on a procedure to control for multiple comparisons which is described in Section 3.15.4.

A comprehensive set of data listings including all randomized subjects will be provided. These listings will include both measured and derived values. Observations in data listings will typically be sorted by subject and timepoint (if applicable).

The derived variable "study day" is used in a number of calculations for data summaries and listings. This variable is calculated as the number of days after a subject's Day -1 visit. Study Day 1, then, is the day after the Day -1 visit.

Summary statistics will be presented using a significant figure rule: the median, minimum, and maximum will have the same number of significant figures as the data; the mean will have one more significant figure than the data being summarized; the SD and SEM will have the same number of significant figures as the mean; and the sample size (N) will be reported as an integer. This rule may be modified if warranted, based on practical considerations.

All analyses, tables, figures, and listings will be generated using SAS® software (version 9.3 or later), unless stated otherwise.

# **3.2.** Sample Size Calculation

The protocol-specified sample size of 30 subjects per treatment group is based on a power calculation for the TTS change from baseline using a two-sample t-test with a two-sided Type I error of 0.05. This sample size provides approximately 80% power to detect an effect size of 0.75 and approximately 90% power to detect an effect size of 0.85. Note that the effect size is defined as the mean difference between an NBI-98854 treatment group and the placebo group

divided by the common SD (eg, a mean difference of 8 divided by an SD of 10 yields an effect size of 0.8).

Standard deviations reported in the literature for TS studies evaluating changes in the TTS (with or without placebo controls) have generally been in the range of 7.5 to 9.5, and in placebo-controlled studies, mean differences between active and placebo arms have been in the range of 5 to 9 (Jankovic et al., 2010; Yoo et al., 2013; ClinicalTrials.gov NCT01727700). The effect sizes of 0.75 and 0.85 mentioned in the above paragraph are representative of effect sizes seen in these published reports.

# 3.3. Pooling of Sites

Approximately 40 study centers are expected to participate in the study. With the exception of the summary of subject enrollment by site, study sites will be pooled in all analyses, tables, and figures, since the majority of sites in this study are of a relatively small size, with fewer than five subjects expected to be enrolled. In addition, study site will not be included as a factor in any statistical models.

# 3.4. Handling of Early Termination Visit Data

An early termination (ET) visit occurs when a subject withdraws from the study prior to completing the scheduled Week 10 visit. An ET visit will be mapped to the next scheduled study visit if it occurs within 7 days prior to and 6 days after the expected study day of the next scheduled visit (with the requirement that the scheduled visit prior to the ET visit was actually completed by the subject). An ET visit at Day 63 or later will be mapped to the Week 10 visit. Early termination visit data which are not mapped to a scheduled visit will be displayed in applicable by-subject data listings but not included in by-visit analyses and summaries.

Table 1 displays the allowable study day range for each scheduled visit for ET visit mapping purposes.

| Scheduled Visit | Target Study Day | Time Interval<br>(Study Day Range) |
|-----------------|------------------|------------------------------------|
| Week 2 | 14 | 7-20 |
| Week 4 | 28 | 21-34 |
| Week 6 | 42 | 35-48 |
| Week 8 | 56 | 49-62 |
| Week 10 | 70 | >62 |

Table 1: Allowable Study Day Range for Early Termination Visit Mapping

# 3.5. Handling of Missing Data

Missing values for outcome measures will not be replaced with imputed values except as noted above for the ET visit data mapped to a scheduled visit for summary and analysis purposes. One exception to this is the imputation of missing values for the sensitivity analyses that will be performed in conjunction with the primary efficacy endpoint analysis as described in Section 3.15.5.

Derived scale total scores (eg, the YGTSS TTS score), which are calculated as the sum of the scores of the individual scale items, will be set equal to missing if any of the individual scale item scores are missing.

Special rules for handling missing and incomplete dates are described below.

# 3.5.1. Missing and incomplete dates

Missing and incomplete ("partial") dates for AEs and concomitant medications will be imputed only for the purpose of estimating the date of the event or medication usage in relationship to study treatment; however, all data listings will display the original dates as reported in the database.

The imputation rules for AE start dates are as follows:

- If the date is completely missing, the date will be imputed as the date of the first dose of study drug following randomization on Day -1;
- If only the day component is missing from the date, the date will be imputed as the date of the first dose of study drug if the date is in the same month and year as the first dose of study drug; otherwise, the missing day component will be imputed as the first day of the month;
- If both the day and month components are missing from the date, the date will be imputed as the date of the first dose of study drug if the date is in the same year as the first dose; otherwise, the missing components will be imputed as 01 January;
- If any of the above imputations result in a start date that is later than an existing complete (not imputed) end date for the event, the start date will be set equal to the end date.

The imputation rules for concomitant medication start dates are as follows:

- If the date is completely missing, the date will be imputed as 01 January in the year of the subject's screening vital signs assessment;
- If only the day component is missing from the date, the date will be imputed as the date of the first dose of study drug if the date is in the same month and year as the first dose of study drug; otherwise, the missing day component will be imputed as the first day of the month;
- If both the day and month components are missing from the date, the date will be imputed as the date of the first dose of study drug if the date is in the same year as the first dose; otherwise, the missing components will be imputed as 01 January;
- If any of the above imputations result in a start date which is later than an existing complete (not imputed) medication stop date, the start date will be set equal to the stop date.

# 3.6. Coding Dictionary

Medical history and AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, version 12.0). Prior and concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary.

# 3.7. Analysis Sets

# 3.7.1. Definition of Analysis Sets

Three analysis sets will be defined for this study.

The safety analysis set will include all subjects who are randomized to a treatment group and dispensed study drug, with the following two exclusions: (a) subjects who withdraw from the study and return all previously dispensed study drug with all doses present, and (b) subjects who have no postbaseline safety data collected. The safety analysis set will be used for all summaries of safety data (eg, AEs and clinical laboratory data) and pharmacokinetic plasma concentration data. Subjects who are dispensed the incorrect treatment at the time of randomization, and remain on the same incorrect treatment during the study will be assigned to the treatment actually received in all summary tables and figures. Subjects who are dispensed a combination of correct and incorrect treatments during the study will be assigned to the randomized treatment in all summary tables and figures.

The primary efficacy analysis set is the intent-to-treat (ITT) analysis set, which will include all subjects in the safety analysis set who have at least one post-randomization TTS value reported at a scheduled visit or mapped ET visit during the 8-week treatment period. The ITT analysis set will be used for summaries and analyses of efficacy data. Treatment group assignment for all summaries and analyses using the ITT analysis set will be based on the randomization schedule.

The per-protocol (PP) analysis set will include all subjects in the ITT analysis set who have a TTS value for the Week 8 visit (including an ET visit mapped to Week 8), have no efficacy-related important protocol deviations (IPDs; described in Section 3.9) and, for subjects in the NBI-98854 treatment groups, have a detectable plasma level of NBI-98854 at the Week 8 visit, a measure of treatment adherence. The PP analysis set will be used for supportive summaries and analyses of the efficacy data. Treatment group assignment for the PP analysis set will follow the rules described above for the safety analysis set.

# 3.7.2. Summary of Analysis Sets

A summary of the number and percentage of subjects included in (and excluded from, as applicable) each analysis set will be provided for each treatment group and overall (for all randomized subjects). The number and percentage of subjects excluded from each analysis set by reason for exclusion will also be provided.

# 3.7.3. Application of Analysis Sets

Summaries of subject disposition, enrollment by study site, analysis set inclusion/exclusion status, and IPDs will include all randomized subjects. All other summaries by analysis set are identified in Table 2.

**Table 2:** Data Summaries by Analysis Set

| | Analysis Set | | |
|-----------------------------------------------|--------------|-----|----|
| Data Summary/Analysis | Safety | ITT | PP |
| Demographics | X | X | X |
| Baseline subject characteristics | X | X | X |
| Medical history | X | | |
| Study drug dosing (including dose reductions) | X | X | |
| Pharmacokinetic plasma concentration data | X | | |
| YGTSS | | X | X |
| RTRS | | X | X |
| PUTS | | X | X |
| CGI-Tics-Severity | | X | X |
| CGI-TS-Improvement | | X | X |
| Adverse events | X | | |
| C-SSRS | X | | |
| ESRS-A | X | | |
| SIGH-D-17 | X | | |
| Y-BOCS | X | | |
| Vital signs | X | | |
| Physical examination | X | | |
| Weight | X | | |
| ECGs | X | | |
| Clinical laboratory data | X | | |
| Prior and Concomitant medications | X | | |

# 3.8. Subject Randomization and Disposition

The summary of subject randomization and disposition will display the number of subjects who were randomized to each treatment group, completed the 8-week treatment period (defined as having completed a scheduled Week 8 visit [does not include ET visits mapped to Week 8]), and completed the study (defined as having completed a scheduled Week 10 visit [does not include ET visits mapped to Week 10]). The number of subjects who did not complete the study will be displayed both overall and by reason for discontinuation.

This summary table will also include an "all subjects" column.

A separate summary of randomization by study site will be presented. This summary will display the number of subjects randomized to each treatment group at each site. An "all subjects" column will be included in the table.

An additional table will display the number of subjects in each treatment group who completed each study visit (screening through Week 10; including mapped ET visits). This table will also include an "all subjects" column and will be based on the safety analysis set.

# 3.9. Important Protocol Deviations

Important protocol deviations (IPDs) are protocol deviations that might significantly affect the completeness, accuracy and/or reliability of the study data or that might significantly affect a subject's rights, safety, or well-being. An assessment of IPDs will be performed by a committee

composed of NBI Clinical Development project team members prior to database lock. Important protocol deviations may include, but are not limited to the following:

- Failure to obtain informed consent from the subject prior to performing any study procedures
- Deviations from key inclusion/exclusion criteria
- Use of prohibited concomitant medications
- Error in drug dispensing which results in a subject not receiving intended randomized treatment
- Significant deviation from protocol-specified dosing regimen
- Significant deviations in YGTSS administration

A summary of the number and percentage of subjects with IPDs by deviation category for each treatment group will be provided for all randomized subjects. All protocol deviations captured in the clinical study database will be included in the data listings.

# 3.10. Demographic Data and Baseline Characteristics

Demographic data (age, gender, race, and ethnicity) and baseline characteristics (age at TS diagnosis, baseline value of TTS [certified site rater scores], height, weight, body mass index [BMI], and CYP2D6 genotype status) will be summarized using descriptive statistics and frequency tables. These data will be summarized by treatment group with an additional "all subjects" column in the summary table.

# 3.11. Medical History

Medical history will be summarized in frequency tables (number and percentage of subjects) by MedDRA System Organ Class (SOC) and Preferred Term (PT) for each treatment group.

# **3.12.** Study Drug Dosing Compliance

Study drug dosing compliance is calculated as the ratio of the estimated number of doses taken by a subject to the expected number of doses that should have been taken (given the length of time the subject participated in the study treatment period), and is expressed as a percentage. A subject is classified as being compliant with study drug administration if their calculated value is 80% or greater. The number and percentage of subjects in each treatment group who are compliant will be presented for Weeks 2, 4, 6, and 8, and for the full treatment period.

The number of doses taken by each subject between two consecutive visits will be estimated by calculating the difference between the number of capsules dispensed at the first visit and the number of capsules returned at the subsequent visit (note that the number of doses taken is equal to the number of capsules taken divided by 2, as each dose is to be taken as 2 capsules of study drug per study protocol). If an ET visit occurs between scheduled visits, the ET visit data will be used in the calculation. If a subject fails to return the study drug kit dispensed at the previous visit, it will be assumed that the number of doses taken by the subject is equal to the number of days between visits (inclusive of the day of the second visit; not to exceed the number of doses dispensed), as subjects are expected to take one dose per day. If a subject is lost to follow-up between scheduled visits, their dosing data will be limited to the last visit at which they were present.

The estimated number of doses taken by a subject across all visits during the treatment period is calculated as the sum of the number of doses taken between each consecutive pair of visits during the treatment period.

The expected number of doses that should have been taken by a subject between or across visits is based on the expected number of days the subject should have dosed with study drug during the interval of interest, which in turn is based on the duration of the subject's study participation during the interval (which may be shorter, for example, if the subject withdraws from the study).

The expected number of days of dosing (and hence, expected number of doses that should have been taken) is calculated as the difference between the visit date of the second of the two visits and the study drug kit dispense date at the first of the two visits. Note that the expected number of days of dosing cannot exceed the total number of doses actually dispensed (each study drug kit in this study contains 17 doses of study drug). If an ET visit occurs between scheduled visits, the ET visit date will be used in the calculation. If a subject is lost to follow-up between scheduled visits, they will be excluded from the compliance calculations for all visits occurring after the last visit at which they were present. If a subject has a missed visit but has previously been dispensed an extra study drug kit that would have been dispensed at the missed visit, they will be excluded from the compliance calculations for all visits beginning with the missed visit, but will be included in the overall treatment period calculations described in the next paragraph.

The dosing compliance calculation across all visits during the study treatment period will follow the logic described above, with the expected number of days of dosing being equal to the difference between the Week 8 (or ET) visit date and the study drug kit dispense date for the Day -1 visit. The estimated number of doses taken by a subject across all visits during the study is calculated as the sum of the number of doses taken between each consecutive pair of visits during the treatment period. If a subject is lost to follow-up prior to Week 8, their dosing compliance will be based on the last study visit at which they were present.

# 3.13. Dose Reduction Summary

The dose reduction summary will present the number and percentage of subjects with a dose reduction for each treatment group at Weeks 2, 4, and 6. Dose reductions at unscheduled visits prior to Week 6 will be included in the summary for the next scheduled visit (ie, Week 2, 4, or 6). Dose reductions at unscheduled visits after Week 6 will be summarized as "After Week 6" in the table. The table will also include the total number and percentage of subjects with a dose reduction at any time during the study treatment period. Note that this summary includes all reports of dose reductions, including those for the placebo and the NBI-98854 40 mg dose treatment groups (which are not true dose reductions).

### 3.14. Pharmacokinetic Data

The plasma concentrations of NBI-98854 and its active metabolite NBI-98782 will be summarized with descriptive statistics by visit (Weeks 2, 4, 6, 8, and 10) and the most recent NBI-98854 dose received by a subject prior to that visit (this is due to the possibility of a subject having a dose reduction from 80 mg to 40 mg). Note that a subject's treatment group for the Week 10 visit summary will reflect the last dose the subject received during the study treatment period.

This summary will also be generated separately for CYP2D6 poor metabolizers vs. non-poor metabolizers.

Concentrations below the lower limit of quantification (BLQ) will be set equal to zero for all plasma concentration summaries. The lower limits of quantification are as follows: (a) NBI-98854: 1.00 ng/mL and (b) NBI-98782: 0.100 ng/mL.

The following additional descriptive statistics will be included in the plasma concentration summary tables: (a) the number of subjects with plasma concentration values greater than or equal to the lower limit of quantification, (b) the geometric mean, and (c) the geometric coefficient of variation (%).

Plasma concentrations of each PK analyte will be summarized with box plots by NBI-98854 dose level at each visit.

# 3.15. Efficacy Data

# 3.15.1. Efficacy Endpoints

The efficacy endpoints for this study are described in detail in the follow sections of this SAP. An overall summary of the efficacy endpoints is presented below in Table 3.

**Table 3: Efficacy Endpoints and Classification** 

| Efficacy Endpoint | <b>Endpoint Classification</b> |
|---|---|
| YGTSS Total Tic Score (TTS) mean change from baseline to Week 8 | Primary |
| CGI-TS-Improvement mean score at Week 8 | Key secondary |
| Percentage of subjects classified as YGTSS TTS responders at Week 8 | Secondary |
| YGTSS Impairment score mean change from baseline to Week 8 | Secondary |
| YGTSS Global Tic Severity score mean change from baseline to Week 8 | Secondary |
| Rush Video-based Tic Rating Scale (RTRS) total score mean change from baseline to Week 8 | Secondary |
| Premonitory Urge for Tics Scale (PUTS) total score mean change from baseline to Week 8 | Secondary |
| CGI-Tics-Severity score mean change from baseline to Week 8 | Secondary |
| Percentage of subjects classified as CGI-TS-Improvement responders at Week 8 | Secondary |
| YGTSS Total Tic Score (TTS) mean change from baseline to Weeks 2, 4, and 6 | Exploratory |
| CGI-TS-Improvement mean score at Weeks 2, 4, and 6 | Exploratory |
| Percentage of subjects classified as YGTSS TTS responders at Weeks 2, 4, and 6 | Exploratory |
| YGTSS Impairment score mean change from baseline to Weeks 2, 4, and 6 | Exploratory |
| YGTSS Global Tic Severity score mean change from baseline to Weeks 2, 4, and 6 | Exploratory |
| Rush Video-based Tic Rating Scale (RTRS) total score mean change from baseline to Weeks 2, 4, and 6 | Exploratory |
| Premonitory Urge for Tics Scale (PUTS) total score mean change from baseline to Weeks 2, 4, and 6 | Exploratory |
| CGI-Tics-Severity score mean change from baseline to Weeks 2, 4, and 6 | Exploratory |
| Percentage of subjects classified as CGI-TS-Improvement responders at Weeks 2, 4, and 6 | Exploratory |

# 3.15.2. Primary Efficacy Endpoint

The primary efficacy endpoint for this study is the mean change from baseline (Day -1) to Week 8 in the YGTSS TTS (Total Tic Score) based on the certified site rater scores. Mean changes from baseline to Weeks 2, 4, and 6 are exploratory efficacy endpoints.

The TTS is defined as the sum of the YGTSS motor tic severity score and phonic (vocal) tic severity score. The motor tic severity score is calculated as the sum of the scores for the 5 motor tic items (number, frequency, intensity, complexity, and interference). The score for each item can range from 0 to 5, for a maximum total score of 25. The vocal (phonic) tic severity score is

calculated similarly. If any one of the 5 items for the motor or vocal tic severity score is not scored (ie, has a missing value), the associated severity score will be set equal to missing. If any of these items has a missing value at a given subject visit, the TTS value for the subject visit will be set equal to missing as well. The TTS value can range from 0 to 50.

Descriptive statistics will be presented by treatment group for the TTS observed values (ie, the raw data) and changes from baseline (Day -1) at each visit from screening through Week 10. Descriptive statistics will be presented for both the ITT and the PP analysis sets.

The primary efficacy endpoint method of analysis will be a mixed-effect model repeated measures (MMRM) analysis, which includes the changes from baseline at Weeks 2, 4, 6, and 8, and is based on the ITT analysis set. The model will include the baseline TTS as a covariate, and treatment group, visit (Week 2, 4, 6, or 8), treatment group by visit interaction, and baseline covariate by visit interaction as fixed effects. Subject will be included as a random effect. Study site will not be included in the model, as there is a large number of sites, with most sites enrolling a small number of subjects.

Treatment group comparisons for each NBI-98854 treatment group vs. placebo at each visit (ie, Weeks 2, 4, 6, and 8) will be performed by constructing linear contrasts (or equivalent program coding) for differences between treatment group least-squares (LS) means. Nominal two-sided p-values for testing the significance of these differences and associated 95% confidence intervals will be reported in summary tables; however, interpretation of the p-values for the two active treatment group comparisons to placebo at Week 8 will be based on the fixed-sequence testing procedure described below in Section 3.15.4.

A supportive analysis using the MMRM model will be performed with the PP analysis set.

The MMRM analysis will be implemented with the PROC MIXED procedure of SAS®, using the restricted maximum likelihood method, an unstructured within-subject covariance matrix, and denominator degrees of freedom from the Kenward-Roger method. In the event that convergence is not obtained with the unstructured covariance matrix, a Toeplitz covariance structure will be used.

An additional supportive analysis of the TTS change from baseline to Week 8 will be performed using an ANCOVA model. The ANCOVA model will include the baseline TTS as a covariate and treatment group as a fixed effect. This analysis will be performed using both the ITT and PP analysis sets.

Mean (±SEM) values of the TTS values at each visit (Day -1 through Week 10) will be summarized in line graphs by treatment group. Similar graphs will be presented for the changes from baseline (Day -1). These graphs will be based on the ITT analysis set.

The LS means (±SEM) from the MMRM analysis will be summarized in line graphs by treatment group for both the ITT and PP analysis sets.

An additional graph will be presented for the TTS changes from baseline to Week 8. This will be a display of the empirical distribution function for each treatment group, and will be based on the ITT analysis set.

# 3.15.3. Key Secondary Efficacy Endpoint

The key secondary efficacy endpoint for this study is the CGI-TS-Improvement mean score at Week 8. Mean scores at Weeks 2, 4, and 6 are exploratory efficacy endpoints.

Each of the CGI-TS-Improvement response categories will be assigned a numerical score as follows:

Very much improved = 1 Much improved = 2 Minimally improved = 3 Not changed = 4 Minimally worse = 5 Much worse = 6 Very much worse = 7

Descriptive statistics (including both categorical variable statistics [using response categories] and continuous variable statistics [using numerical scores]) will be presented by treatment group for the CGI-TS-Improvement data at each visit from Week 2 through Week 10. Descriptive statistics will be presented for both the ITT and the PP analysis sets.

An analysis of the CGI-TS-Improvement numerical scores at Week 8 will be performed using an ANOVA model which includes treatment group as a fixed effect. The Week 2, 4, and 6 data will be analyzed also using the same ANOVA model. Nominal two-sided p-values for testing the significance of the mean difference between each NBI-98854 treatment group and the placebo group and associated 95% confidence intervals will be reported in summary tables; however, interpretation of the p-values for the two active treatment group comparisons to placebo at Week 8 will be based on the fixed-sequence testing procedure described below in Section 3.15.4.

Supportive analyses of the CGI-TS-Improvement numerical scores will be performed using an ANOVA at each visit based on the PP analysis set.

Mean (±SEM) values of the CGI-TS-Improvement numerical scores at each visit will be summarized in line graphs by treatment group. These graphs will be based on the ITT analysis set.

The LS means (±SEM) from the ANOVA analyses of the CGI-TS-Improvement numerical scores at Weeks 2 through 8 will be summarized in line graphs by treatment group for both the ITT and PP analysis sets.

### 3.15.4. Fixed-Sequence Testing Procedure to Control for Multiple Comparisons

A fixed-sequence testing procedure will be followed for the primary and key secondary efficacy endpoint analyses in order to control for multiple comparisons (ie, comparing each of the two NBI-98854 doses to placebo for each of the two endpoints). The fixed-sequence testing procedure will consist of performing the hypothesis tests in the following pre-specified order:

- Week 8 TTS mean change from baseline: NBI-98854 80 mg treatment group vs. placebo treatment group
- Week 8 TTS mean change from baseline: NBI-98854 40 mg treatment group vs. placebo treatment group

- Week 8 CGI-TS-Improvement mean score: NBI-98854 80 mg treatment group vs. placebo treatment group
- Week 8 CGI-TS-Improvement mean score: NBI-98854 40 mg treatment group vs. placebo treatment group

In order for a test result in the above list to be considered statistically significant, all of the test results higher in the list must be significant at the 0.05 level of significance.

# 3.15.5. Sensitivity Analyses for Primary Efficacy Endpoint

An underlying assumption of the MMRM analysis is that missing data are considered to be missing at random (MAR). In addition to assessing the number of subjects who prematurely discontinue from the study prior to Week 8 along with the reasons for premature study discontinuation, three sensitivity analyses of the TTS changes from baseline will be performed to assess the impact of deviations from the assumption that the missing TTS data are MAR. These analyses, described below, are based on the ITT analysis set.

Tipping Point - Sensitivity Analysis #1

# Step 1 of Sensitivity Analysis #1 (Imputation of Missing Data)

The initial step will be to impute missing TTS values at Weeks 2 through 8 using the SAS® procedure PROC MI. The data will first be examined to determine if the pattern of missing data is monotone or non-monotone across visits from Day -1 (baseline) through Week 8. If the pattern of missing data is monotone (which will be the case if the missingness is purely due to dropouts) the regression method of PROC MI will be used to impute the missing data. If the pattern of missing data is non-monotone, the Markov chain Monte Carlo (MCMC) method of PROC MI will be used to create a monotone data set, using default system values for the parameters CHAIN, NBITER and NITER (along with IMPUTE=MONOTONE). This data set can then be analyzed using the regression method of PROC MI. In either case, 100 imputed data sets will be generated using a random number generator seed value of 1470681. The SAS® statements (or equivalent) provided below will be used for the imputation of missing data. Note that "Treat" represents randomized treatment group (placebo, NBI-98854 40 mg, or NBI-98854 80 mg), "Baseline" is the Day -1 TTS value, and Week2, Week4, Week6, and Week8 are the TTS values at Weeks 2, 4, 6, and 8, respectively.

PROC MI NIMPUTE=100 SEED=1470681 MINIMUM=0 MAXIMUM=50 OUT=Imputed; CLASS Treat; MONOTONE REGRESSION; VAR Treat Baseline Week2 Week4 Week6 Week8;

# <u>Step 2 of Sensitivity Analysis #1 (Creation of Additional Data Sets with NBI-98854 Treatment</u> Group Imputed TTS Scores Made Worse in a Step-Wise Fashion)

The sensitivity analysis itself will involve the creation of additional data sets based on the fully imputed data sets created in Step 1, with a step-wise "worsening-score" algorithm applied to the NBI-98854 treatment groups, but not to the placebo treatment group. Since the primary endpoint is the TTS mean change from baseline at Week 8, the scores at Weeks 2, 4, and 6, which were used for missing data imputation purposes, will not be used in any subsequent calculations or analyses. Therefore, the worsening-score algorithm will be applied only to the NBI-98854

treatment group imputed Week 8 TTS values (also note that the method of analysis for the imputed data sets described below in Step 3 is an ANCOVA of the Week 8 TTS changes from baseline).

The worsening-score algorithm will involve increasing (or "worsening") the imputed Week 8 TTS values in the two NBI-98854 treatment groups by a percentage of the imputed value in a pre-specified, step-wise fashion. Imputed Week 8 TTS values in the placebo treatment group will not be made worse in this algorithm and will remain at the initially imputed values.

The initial percentage value to be applied is 10%. This will be increased in fixed increments of 10% until the p-value for the comparison of the NBI-98854 80 mg treatment group to the placebo treatment group (obtained as described below in Step 3 from PROC MIANALYZE applied to the results of 100 ANCOVAs for each imputed data set) exceeds the nominal 0.05 level of significance. Note that the maximum possible value for the TTS is 50; therefore an imputed Week 8 TTS value adjusted according to this algorithm cannot exceed the value of 50.

This sensitivity analysis represents a tipping point analysis based on "delta adjustments," which is a commonly used approach to assess the impact of missing data in clinical trials (O'Kelly and Ratitch, 2014).

# Step 3 of Sensitivity Analysis #1

The TTS changes from baseline to Week 8 will be calculated for each of the imputed data sets from the original PROC MI output and for the additional sets of data created according to the worsened-score algorithm described above in Step 2. The imputed data sets will be analyzed using the ANCOVA model specified above in Section 3.15.2, using either PROC MIXED or PROC GLM.

PROC MIANALYZE will then be used to combine results from the 100 ANCOVAs for the imputed data sets to provide the following statistics:

- LS mean for each treatment group
- LS mean difference between each NBI-98854 treatment group and the placebo treatment group, along with the corresponding two-sided 95% confidence intervals and p-values

# Jump to Reference (J2R) - Sensitivity Analysis #2

The J2R method is based on the concept that missing values for subjects in the NBI-98854 treatment groups who drop out prior to the Week 8 visit will tend to be similar to values for subjects in the reference (placebo) group who have similar baseline characteristics. This is plausible under the assumption that treatment with NBI-98854 offers symptomatic, and not disease-modifying treatment, and as such, subjects who stop taking active study drug will no longer benefit from its therapeutic effect, but will still be subject to any placebo (or study participation related) effects.

The J2R analysis will be implemented using the SAS® procedures PROC MI and PROC MIANALYZE. If the pattern of missing data across study visits during the treatment period is non-monotone, a monotone data set will be created using PROC MI with the MCMC method, a seed value of 1470681, and system default values for the parameters CHAIN, NBITER, and NITER (along with IMPUTE=MONOTONE). The number of imputed data sets created in this step will be 100.

The actual J2R imputation will follow the sequential model approach described in Chapter 7.4.3 of O'Kelly and Ratitch (2014). With this approach, the placebo treatment group data are used to impute missing values for the NBI-98854 treatment groups, one visit at a time in a sequential fashion. At each visit imputation step, PROC MI with the same seed specified in the preceding paragraph (and 100 imputed data sets) will be implemented, using the monotone regression method with the baseline TTS as an explanatory variable. Note that missing data values in the placebo treatment group are imputed under the MAR assumption (using PROC MI with the monotone regression method), prior to imputing missing data values in the NBI-98854 treatment groups.

The final step of this analysis will consist of performing an ANCOVA analysis of the TTS changes from baseline at Week 8 using the imputed data sets and then combining the results of these analyses using PROC MIANALYZE.

# Baseline Observation Carried Forward (BOCF) – Sensitivity Analysis #3

The use of a BOCF analysis as a sensitivity analysis is described in a publication authored by Dr. Lisa LaVange of the FDA/CDER Office of Biostatistics (LaVange, 2014). This analysis will be implemented by imputing missing Week 8 TTS values in all three treatment groups with the baseline values (ie, a subject's missing Week 8 value will be set equal to their baseline value). The TTS changes from baseline at Week 8, including BOCF-imputed missing values for Week 8, will then be analyzed using the ANCOVA model, using either PROC MIXED or PROC GLM. As this is a single-imputation method, the use of PROC MI and PROC MIANALYZE is not required.

# 3.15.6. Secondary Efficacy Endpoints

#### 3.15.6.1. YGTSS TTS Responder Analysis

A TTS responder is defined, on a per-visit basis, as a subject whose TTS value is reduced by at least 30% from baseline (Day -1) at the specified postbaseline visit. The percentage of subjects classified as TTS responders will be summarized for each treatment group at Weeks 2, 4, 6, 8, and 10 for both the ITT and PP analysis sets.

The percentage of subjects classified as TTS responders at Week 8 is a secondary efficacy endpoint. An analysis comparing each NBI-98854 treatment group to the placebo treatment group will be performed for this endpoint with the ITT analysis set using the standard chi-square test. A separate chi-square test will be performed for each treatment group comparison (NBI-98854 80 mg treatment group vs. placebo treatment group and NBI-98854 40 mg treatment group vs. placebo treatment group).

A supportive analysis of the percentage of subjects classified as TTS responders at Week 8 will be performed using the PP analysis set.

The percentages of subjects classified as TTS responders at Weeks 2, 4, and 6 are exploratory endpoints. These endpoints will be analyzed using the chi-square test at each of these visits with both the ITT and PP analysis sets.

Bar graphs displaying the percentage of subjects classified as TTS responders will be presented by treatment group for each study visit from Week 2 through Week 10 for the ITT and PP analysis sets.

# 3.15.6.2. YGTSS Impairment Score

The YGTSS Impairment score can range in value from 0 to 50. The YGTSS Impairment score mean change from baseline to Week 8 is a secondary efficacy endpoint. Mean changes from baseline to Weeks 2, 4, and 6 are exploratory efficacy endpoints.

Descriptive statistics will be presented by treatment group for the YGTSS Impairment score observed values (ie, the raw data) and changes from baseline (Day -1) at each visit from screening through Week 10. Descriptive statistics will be presented for both the ITT and the PP analysis sets.

The analysis of the YGTSS Impairment score changes from baseline at each visit from Week 2 through Week 8 will be performed using a MMRM model similar to the model described in Section 3.15.2 for the TTS change from baseline, based on the ITT analysis set. The covariate for this MMRM model will be the YGTSS Impairment score at baseline. A supportive analysis of the YGTSS Impairment score changes from baseline will be performed using the PP analysis.

Mean (±SEM) values of the YGTSS Impairment score at each visit (Day -1 through Week 10) will be summarized in line graphs by treatment group. Similar graphs will be presented for the changes from baseline (Day -1). These graphs will be based on the ITT analysis set.

The LS means (±SEM) from the MMRM analysis of the YGTSS Impairment score changes from baseline will be summarized in line graphs by treatment group for both the ITT and PP analysis sets.

# 3.15.6.3. YGTSS Global Tic Severity Score

The YGTSS Global Tic Severity score is the sum of the TTS and the YGTSS Impairment score. The YGTSS Global Tic Severity score at a given subject visit will be set equal to missing if either of the TTS or Impairment scores are missing. The YGTSS Global Tic Severity score value can range from 0 to 100.

The YGTSS Global Tic Severity score mean change from baseline to Week 8 is a secondary efficacy endpoint. Mean changes from baseline to Weeks 2, 4, and 6 are exploratory efficacy endpoints.

Descriptive statistics will be presented by treatment group for the YGTSS Global Tic Severity score observed values (ie, the raw data) and changes from baseline (Day -1) at each visit from screening through Week 10. Descriptive statistics will be presented for both the ITT and the PP analysis sets.

An analysis of the YGTSS Global Tic Severity change-from-baseline scores at each visit from Week 2 through Week 8 will be performed using a MMRM model similar to the model described in Section 3.15.2 for the TTS change from baseline, based on the ITT analysis set. The covariate for this MMRM model will be the YGTSS Global Tic Severity score at baseline. A supportive analysis of the YGTSS Global Tic Severity scores will be performed using the PP analysis set.

Mean (±SEM) values of the YGTSS Global Tic Severity score at each visit (Day -1 through Week 10) will be summarized in line graphs by treatment group. Similar graphs will be presented for the changes from baseline (Day -1). These graphs will be based on the ITT analysis set.

The LS means (±SEM) from the MMRM analysis of the YGTSS Global Tic Severity score changes from baseline will be summarized in line graphs by treatment group for both the ITT and PP analysis sets.

# 3.15.6.4. Rush Video-based Tic Rating Scale (RTRS)

The modified RTRS used in this study includes short video recordings to measure 5 tic variables: number of body areas affected, frequency of motor and phonic tics, and severity of motor and phonic tics. The RTRS videos for Day -1 and Week 8 (or final on-treatment visit for subjects who discontinue from the study prior to Week 8) will be reviewed and scored by a pair of blinded central raters using a consensus scoring process that is blinded to both treatment and visit sequence. The summaries and analyses of the RTRS data, then, will be limited to the scores recorded for these two visits for each subject.

The RTRS total score is calculated as the sum of the 5 domain scores (number of body areas affected, motor tic frequency, phonic tic frequency, severity of motor tics, and severity of phonic tics). The score for each domain can range from 0 to 4, for a maximum possible total score of 20. If any one of the 5 domains is not scored (ie, has a missing value), the total score will be set equal to missing.

The RTRS total score mean change from baseline to Week 8 (or final on-treatment visit if prior to Week 8) is a secondary efficacy endpoint.

Descriptive statistics will be presented by treatment group for the RTRS total score observed values (ie, the raw data) at each visit and changes from baseline (Day -1). Descriptive statistics will be presented for both the ITT and the PP analysis sets.

An analysis of the RTRS total score changes from baseline to Week 8 (or final on-treatment visit if prior to Week 8) will be performed using an ANCOVA model similar to the model described in Section 3.15.2 for the TTS change from baseline. The covariate for this analysis will be the RTRS total score at baseline. A supportive analysis of the RTRS total scores will be performed using the PP analysis set.

Mean (±SEM) values of the RTRS total score for each treatment group at each visit will be summarized in a bar graph. A similar graph will be presented for the changes from baseline. These graphs will be based on the ITT analysis set.

The LS means (±SEM) from the ANCOVA analysis of the RTRS total score changes from baseline to Week 8 (or final on-treatment visit if prior to Week 8) will be summarized in a bar graph by treatment group for both the ITT and PP analysis sets.

# 3.15.6.5. Premonitory Urge for Tics Scale (PUTS)

The PUTS consists of 9 items, each of which is scored on a 4-point scale (1=not at all true, 2=a little true, 3=pretty much true, 4=very much true). The PUTS total score is calculated as the sum of the scores for the 9 items. The maximum possible total score is 36. If any one of the 9 items is not scored (ie, has a missing value), the PUTS total score will be set equal to missing.

The PUTS total score mean change from baseline to Week 8 is a secondary efficacy endpoint. Mean changes from baseline to Weeks 2, 4, and 6 are exploratory efficacy endpoints.

Descriptive statistics will be presented by treatment group for the PUTS total score observed values (ie, the raw data) and changes from baseline (Day -1) at each visit from screening through Week 10. Descriptive statistics will be presented for both the ITT and the PP analysis sets.

An analysis of the PUTS total score changes from baseline at each visit from Week 2 through Week 8 will be performed using a MMRM model similar to the model described in Section 3.15.2 for the TTS change from baseline. The covariate for this MMRM analysis will be the PUTS total score at baseline. A supportive analysis of the PUTS total scores will be performed using the PP analysis set.

Mean (±SEM) values of the PUTS total score at each visit (Day -1 through Week 10) will be summarized in line graphs by treatment group. Similar graphs will be presented for the changes from baseline. These graphs will be based on the ITT analysis set.

The LS means (±SEM) from the MMRM analysis of the PUTS total score changes from baseline to Weeks 2 through 8 will be summarized in line graphs by treatment group for both the ITT and PP analysis sets.

# 3.15.6.6. CGI-Tics-Severity

Each of the CGI-Tics-Severity response categories will be assigned a numerical score as follows:

- Normal, not at all ill = 1
- Borderline ill = 2
- Mildly ill = 3
- Moderately ill = 4
- Markedly ill = 5
- Severely ill = 6
- Among the most extremely ill patient = 7

The CGI-Tics-Severity numerical score mean change from baseline to Week 8 is a secondary efficacy endpoint. Mean changes from baseline to Weeks 2, 4, and 6 are exploratory efficacy endpoints.

Descriptive statistics (including both categorical variable statistics [using response categories] and continuous variable statistics [using numerical scores]) will be presented by treatment group for the CGI-Tics-Severity data at each visit from screening through Week 10. Changes from baseline (Day -1) for the numerical scores will be summarized also. Descriptive statistics will be presented for both the ITT and the PP analysis sets.

An analysis of the CGI-Tics-Severity numerical score changes from baseline to each visit from Week 2 through Week 8 will be performed using a MMRM model similar to the model described in Section 3.15.2 for the TTS changes from baseline. The covariate for this MMRM analysis will be the CGI-Tics-Severity numerical score at baseline. A supportive analysis of the CGI-Tics-Severity numerical scores will be performed using the PP analysis set.

Mean (±SEM) values of the CGI-Tics-Severity numerical scores at each visit (Day -1 through Week 10) will be summarized in line graphs by treatment group. Similar graphs will be presented for the changes from baseline. These graphs will be based on the ITT analysis set.

The LS means (±SEM) from the MMRM analysis of the CGI-Tic-Severity numerical score changes from baseline to Weeks 2 through 8 will be summarized in line graphs by treatment group for both the ITT and PP analysis sets.

# 3.15.6.7. CGI-TS-Improvement Responder Analysis

A subject is classified as a CGI-TS-Improvement responder at a given visit if their CGI-TS-Improvement score is either a "1" ("very much improved") or a "2" ("much improved") at the visit.

The percentage of subjects classified as CGI-TS-Improvement responders at Week 8 is a secondary efficacy endpoint. The percentages of responders at Weeks 2, 4, and 6 are exploratory efficacy endpoints.

The number and percentage of responders will be summarized for each treatment group at Weeks 2, 4, 6, 8, and 10. The CGI-TS-Improvement responder summary statistics will be presented for both the ITT and the PP analysis sets.

An analysis comparing each NBI-98854 treatment group to the placebo treatment group will be performed for the percentage of subjects classified as CGI-TS-Improvement responders at each of Weeks 2 through 8 using the standard chi-square test with the ITT analysis set. A separate chi-square test will be performed for each NBI-98854 treatment group comparison to placebo for each visit.

A supportive analysis of the percentage of subjects classified as CGI-TS-Improvement responders at Weeks 2 through 8 will be performed using the PP analysis set.

Bar graphs displaying the percentage of subjects classified as CGI-TS-Improvement responders at Weeks 2 through 10 will be presented by treatment group for the ITT and the PP analysis sets.

# 3.16. Safety Data

#### 3.16.1. Adverse Events

A treatment-emergent adverse event (TEAE) is any reaction, side effect, or other untoward event, regardless of relationship to study drug, that is newly reported or considered a worsening or change in nature, severity, or frequency of conditions present at the start of the study which occurs any time after first dose of study drug.

TEAEs, categorized by MedDRA (Version 12.0) system organ class (SOC) and preferred term (PT), will be summarized by treatment group in frequency tables. Each table will also include a separate column for all NBI-98854 treated subjects (ie, excluding placebo subjects). Unless stated otherwise, the frequency tables will include the number of events reported, and the number and percentage of unique subjects experiencing each event one or more times during the study. SOCs will be displayed in order of decreasing frequency (number of subjects with TEAEs in the SOC based on the "all NBI-98854 treated subjects" column), and within each SOC, PTs will be displayed in a similar fashion in order of decreasing frequency of subjects with TEAEs in the PT based on the "all NBI-98854 treated subjects" column.

Two versions of the primary TEAE frequency table will be presented: (a) the first version as described above which includes both SOC and PT, with each sorted in decreasing frequency based on the "all NBI-98854 treated subjects" column, and (b) a second version which does not

include SOCs but does include PTs sorted in decreasing frequency based on the "all NBI-98854 treated subjects" column.

Frequency tables will be presented including only TEAEs considered to be possibly or definitely related to study drug and categorizing TEAEs according to the maximum intensity reported for a given subject.

AEs with an onset date during screening (prior to study drug dosing) will be presented only in a data listing.

## 3.16.1.1. Adverse Event Overall Summary

An overall summary table will be provided which summarizes the number and percentage of subjects in each treatment group with any TEAE, any treatment-related TEAE (ie, possibly or definitely related), any severe TEAE, any TEAE leading to dose reduction, any TEAE leading to study discontinuation, any serious TEAE, and any TEAE resulting in death.

#### 3.16.1.2. Adverse Events Resulting in Study Drug Dose Reductions

A summary table of TEAEs resulting in study drug dose reductions will be presented. The first line of the table will display the overall frequency for each treatment group column. Note that subjects randomized to the placebo and NBI-98854 40 mg treatment groups who have a reported dose reduction actually remain on the randomized dose, while subjects randomized to the NBI-98854 80 mg treatment group will have an actual dose reduction.

A listing of TEAEs resulting in a study drug dose reduction will be provided. This listing will include subject, treatment group, study day of the dose reduction, and additional information from the AE eCRF.

## 3.16.1.3. Adverse Events Resulting in Premature Study Discontinuation

A summary table of TEAEs resulting in premature study discontinuation will be presented. The first line of the table will display the overall frequency for each treatment group column.

A listing of TEAEs resulting in premature study discontinuation will be included in the study report as a table. The listing will include subject, treatment group, last treatment received prior to the onset time of the TEAE leading to discontinuation, study day of the discontinuation, and both the PT and reported (verbatim) term for all TEAEs that resulted in the premature study discontinuation.

#### 3.16.1.4. Deaths and Other Serious Adverse Events

The frequency of serious adverse events (SAEs) will be summarized using the approach described in Section 3.16.1.3. The table format for the SAE tables will match those used for the TEAE discontinuation tables. Deaths will be presented in a listing only.

Listings of SAEs and deaths will be provided. These listings will include subject, treatment group, last treatment received prior to the onset time of the SAE or the TEAE leading to death, study day of the death or SAE onset, and all other AE-specific information reported on the AE eCRF.

# 3.16.2. Clinical Laboratory Data

The hematology, clinical chemistry, and prolactin data will be summarized with descriptive statistics by treatment group at each scheduled visit from screening (from Day -1 for prolactin) through Week 10. Both observed values and changes from baseline (Day -1, or screening if the Day -1 value is missing) will be summarized.

The prolactin data will be summarized by visit and treatment group for each gender separately, in addition to the summaries described above.

Shift tables will be presented for selected clinical laboratory variables based on the reference range-based categories of "Low," "Normal," or "High." An observed clinical laboratory variable value will be assigned to one of these three categories according to the reference ranges provided by the central clinical laboratory.

Each shift table will have three rows and three columns, with rows reflecting the reference range category at baseline, and columns reflecting the reference range category at Week 8. Subjects with missing data for a clinical laboratory variable at either baseline or at Week 8 will not be included in the table for that variable. The number and percentage of subjects in each shift category will be displayed in the table.

Shift tables will be presented for the following clinical laboratory variables: aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), total bilirubin, creatine kinase, creatinine, blood urea nitrogen, prolactin, white blood cell count, absolute neutrophil count, hemoglobin, and platelet count.

Summaries of sponsor-defined potentially clinically significant (PCS) values will be presented for the following clinical laboratory variables: ALT, AST, creatinine kinase, GGT, total bilirubin, white blood cell count, absolute neutrophil count, creatinine, and BUN. The number and percentage of subjects with PCS values that are reported at any postbaseline visit (scheduled or unscheduled) will be summarized by treatment group in summary tables. The criteria for identifying PCS clinical laboratory values are provided in Table 4.

**Table 4: Potential Clinically Significant Criteria for Clinical Laboratory Variables** 

| Variable | PCS Threshold |
|---------------------------|------------------------------------|
| ALT | >3 x ULN (upper limit of normal) |
| AST | >3 x ULN |
| Creatine kinase | >5 x ULN |
| GGT | >3 x ULN |
| Total bilirubin | >1.5 x ULN |
| White blood cell count | ≤2.8 x 1000/μL |
| Absolute neutrophil count | <1.5 x 1000/μL |
| Creatinine | >1.5 x Day -1 value or > 1.5 x ULN |
| BUN | >30 mg/dL (> 10.71 mmol/L) |

A listing of subjects with PCS values at any postbaseline visits for any of the variables listed in the table above will be presented. The listing will include subject, treatment group, visit, study day, and, for each subject, all laboratory results (including all scheduled and unscheduled visits) for the variables with a PCS value for that subject. Values that meet the PCS criteria will be flagged with an asterisk in the listing.

Scatter plots of selected variables will be created which display Week 8 values vs. baseline values. Each plot will include a 45 degree ("y=x") reference line. The plots will be generated by treatment group for ALT, AST, creatine kinase, GGT, total bilirubin, and prolactin.

Additional graphs will be presented for the prolactin data. These graphs will display mean (±SEM) prolactin values for each treatment group at each scheduled visit (Day -1 through Week 10) in a line graph layout. A separate graph will be presented for each gender, and each graph will be annotated with the reference range lower and upper limits displayed as horizontal dashed lines.

The clinical laboratory data listings located in Section 16.2 of the study report will include associated reference ranges (if provided). In addition, values outside the reference range will be flagged as "L" if below the lower limit of normal and as "H" if above the upper limit of normal. There will also be a flag for clinical significance based on the investigator's assessment of out-of-range values. The urinalysis data will be presented in data listings only.

Repeat clinical laboratory samples may be collected at any time during this study due to either missing or abnormal results. The general rule for summarizing these data is to include the original sample results in summary tables and graphs. One exception to this rule is when there are missing results from the original samples at screening – in this situation, the results of a repeat screening sample will be substituted for the missing results in summary tables and graphs. All sample results (original and repeat) will be included in data listings.

# 3.16.3. Physical Examination and Weight

Clinically significant physical examination findings will be presented by subject and visit in a listing. The listing will include subject, visit at which the finding was reported, study day, treatment group, and the clinically significant finding.

Body weight, which is measured during the physical examination, will be summarized in units of kilograms with descriptive statistics (both observed values and changes from baseline [Day -1, or screening if the Day -1 value is missing]) by treatment group at each scheduled visit from screening through Week 10.

# **3.16.4. Vital Signs**

The vital signs data, including orthostatic blood pressures and heart rate (calculated as standing value minus supine value), will be summarized with descriptive statistics by treatment group at each scheduled visit from screening through Week 10. Both observed values and changes from baseline (Day -1, or screening if the Day -1 value is missing) will be summarized.

Sponsor-defined PCS values for systolic blood pressure, diastolic blood pressure, and heart rate will be summarized by treatment group. The number and percentage of subjects with PCS values at any postbaseline visit (scheduled or unscheduled) will be presented in the summary tables. The criteria for identifying PCS vital signs values are provided in Table 5.

| Table 5: Potential | ly Clinically Si | gnificant Criteria f | for Vital Signs |
|---|---|---|---|
|---|---|---|---|

| Variable Name | PCS – Low if: | | PCS – High if: | | |
|---|---|---|---|---|---|
| | Observed<br>Value is: AND | Decrease from Baseline is: | Observed Value is: | AND | Increase from Baseline is: |
| Systolic Blood<br>Pressure | <90 mmHg | ≥20 mmHg | >180 mmHg | | ≥20 mmHg |
| Diastolic Blood<br>Pressure | <50 mmHg | ≥10 mmHg | >105 mmHg | | ≥15 mmHg |
| Heart Rate | <50 bpm | ≥15 bpm | >120 bpm | | ≥15 bpm |

Note that both supine and standing values of blood pressures and heart rate at all postbaseline visits will be included in the identification and summary of PCS values.

A listing of vital signs data at all visits (scheduled and unscheduled) for subjects with PCS values will be presented. The listing will include subject, treatment group, visit, study day, systolic blood pressure (supine and standing), diastolic blood pressure (supine and standing), and heart rate (supine and standing). Values that meet the PCS criteria will be flagged with an asterisk in the listing.

# 3.16.5. Electrocardiogram

The triplicate values of the quantitative ECG variables (heart rate, PR interval, QRS duration, QT interval, and Fridericia's correction of QT interval [QTcF]) measured at each visit will be averaged for the purpose of analysis. For the overall assessment categorical variable (the investigator's assessment of the ECG as Normal, Abnormal not Clinically Significant, or

Abnormal Clinically Significant), which is also reported in triplicate, the value that represents the greatest degree of abnormality will be used in all summary tables.

The ECG variables will be summarized with descriptive statistics (frequency tables for the overall assessment categorical variable) by treatment group at each scheduled visit from screening through Week 10. Both observed values and changes from baseline (Day -1, or screening if the Day -1 value is missing) will be summarized (for the overall categorical assessment, only observed values will be summarized).

Categorical summaries will be presented for the QT and QTcF interval data. For these summaries, a subject's highest reported postbaseline value will be used to determine in which category(s) the subject will be counted.

Two categorical summaries will be presented for the QT and QTcF intervals (each interval will be summarized separately). For the first summary, the number and percentage of subjects in each treatment group whose highest reported QT/QTcF postbaseline value meets the following thresholds will be summarized:

- Greater than 450 msec
- Greater than 480 msec
- Greater than 500 msec

The second categorical summary will display the number and percentage of subjects in each treatment group whose largest QT/QTcF increase from their baseline value meets the following thresholds:

- Greater than 30 msec
- Greater than 60 msec

# 3.16.6. Columbia-Suicide Severity Rating Scale (C-SSRS)

The C-SSRS data will be presented in the following summaries:

- Screening/lifetime assessment by treatment group and for all subjects combined
- Screening/past 1 year assessment by treatment group and for all subjects combined
- Baseline (Day -1) assessment by treatment group and for all subjects combined
- All postbaseline assessments (Day 1 through Week 10) by treatment group

Each summary will display the number and percentage of subjects who report "Yes" to specific C-SSRS items or categories of items (a category is assigned a "Yes" value if a "Yes" is reported for any item in the category). These C-SSRS items and categories are as follows:

- Suicidal Ideation Items
  - (1) Wish to be dead
  - (2) Non-specific active suicidal thoughts
  - (3) Active suicidal ideation with any methods (not plan) without intent to act
  - (4) Active suicidal ideation with some intent to act, without specific plan
  - (5) Active suicidal ideation with specific plan and intent

- Suicidal Ideation Category: Any of items (1) through (5)
- Suicidal Behavior Items (not reported for the Screening/past 1 year assessment)
  - (6) Preparatory acts or behavior
  - (7) Aborted attempt
  - (8) Interrupted attempt
  - (9) Non-fatal suicide attempt
  - (10) Completed suicide
- Suicidal Behavior Category: Any of items (6) through (10)
- Suicidal Ideation or Behavior Category: Any of items (1) through (10)

For the "all postbaseline assessments" summary, each subject's C-SSRS responses for all postbaseline assessments during the study (including assessments at both scheduled and unscheduled visits) will be evaluated, and a "Yes" response for any assessment will be considered as a "Yes" for the subject.

In addition to the summaries described above, shift tables comparing postbaseline suicidal ideation scores to baseline scores will be presented. The shift table scores are defined as the following:

- 0=No suicidal ideation
- 1=Wish to be dead
- 2=Non-specific active suicidal thoughts
- 3=Active suicidal ideation with any methods (not plan) without intent to act
- 4=Active suicidal ideation with some intent to act, without specific plan
- 5=Active suicidal ideation with specific plan and intent

The shift tables will display the number and percentage of subjects within each cell of a 6 x 6 table for each treatment group, with the rows representing the baseline score and the columns representing the maximum score recorded across all postbaseline assessments (including both scheduled and unscheduled visits). Subjects missing either a baseline score or all postbaseline scores will not appear in the table.

A summary listing of individual subject data for the C-SSRS will be provided which lists data at all visits for subjects with a positive response for suicidal ideation, suicidal behavior, or self-injurious behavior without suicidal intent at any postbaseline visit during the study. The listing will be in the form of a table, with each row representing a subject visit (scheduled and unscheduled). The listing will include subject, visit, timepoint (for screening assessments), study day of the visit, treatment group, and a column for each suicidal ideation item (1-5), each suicidal behavior item (6-10), and a final column for self-injurious behavior without suicidal intent. The cells of the table will be populated with "Y" or "N," representing either a positive or negative response, respectively, for each item in the table (ie, for each column of the table).

# 3.16.7. Extrapyramidal Symptom Rating Scale-Abbreviated (ESRS-A)

Amendment 3 of the clinical study protocol added the ESRS-A assessment tool to evaluate extrapyramidal symptoms, therefore it is expected that data will be available for all subject visits that take place after the date of the IRB approval at each site.

The ESRS-A assesses 4 types of movement disorders: parkinsonism, dystonia, akathisia, and tardive dyskinesia. The ESRS-A consists of four subscales, one for each type of movement disorder. The ESRS-A contains 10 items to evaluate parkinsonism, 6 items to evaluate dystonia, 6 items to evaluate dyskinesia, and 2 items to evaluate akathisia. Each item score can range from 0 to 5, for a maximum possible parkinsonism score of 50, maximum possible dystonia score of 30, maximum possible dyskinesia score of 30, and maximum possible akathisia score of 10. A Clinical Global Impression of Severity (CGI-S) is also completed for each type of movement disorder, and is also is scored on a 0 to 5 scale. The ESRS-A is administered at baseline (Day -1) and at Weeks 2, 4, 6, 8, and 10.

The subscale scores for each type of movement disorder (parkinsonism, akathisia, dystonia, and tardive dyskinesia) will be calculated as the sum of the scores of the individual items comprising each subscale. The overall total score will be calculated as the sum of each of the subscale scores. If any one of the items is not scored (ie, has a missing value), the associated subscale score and total score will be set equal to missing. The CGI-S scores will be summarized separately from the subscale scores.

Each of the subscale scores for parkinsonism, akathisia, dystonia, and tardive dyskinesia, and the overall total score at each visit (Day -1 and Weeks 2, 4, 6, 8, and 10) will summarized with descriptive statistics by treatment group. Changes from baseline at each post-baseline visit will also be summarized.

The CGI-S scores for each subscale at each visit (Day -1 and Weeks 2, 4, 6, 8, and 10) will summarized with descriptive statistics by treatment group. Changes from baseline at each post-baseline visit will also be summarized.

# 3.16.8. Yale-Brown Obsessive Compulsive Scale (Y-BOCS)

The Y-BOCS is a semi-structured interview designed to rate the severity of obsessive and compulsive symptoms.

The Y-BOCS obsession subtotal score is calculated as the sum of the scores for items 1 through 5 of the Y-BOCS scale (excluding item 1b), and the Y-BOCS compulsion subtotal score is calculated as the sum of the scores for items 6 through 10 of the Y-BOCS scale (excluding item 6b). The Y-BOCS total score is the sum of the obsession and compulsion subtotal scores. Each item score ranges from 0 to 4, with a maximum possible obsession subtotal score of 20, a maximum possible compulsion subtotal score of 20, and a maximum possible total score of 40. If any one of these 10 items is not scored (ie, has a missing value), the associated subtotal score and total score will be set equal to missing.

The subtotal scores for obsession and compulsion, and the total score at each visit (screening, Day -1, and Weeks 2, 4, 6, 8, and 10) will summarized with descriptive statistics by treatment group. Changes from baseline (Day -1) at each postbaseline visit will also be summarized.

# 3.16.9. Structured Interview Guide for the Hamilton Depression Rating Scale (SIGH-D-17)

The SIGH-D-17 is a 17-item, semi-structured questionnaire for rating depression and is administered by the investigator (or designee). The SIGH-D-17 total score is calculated as the sum of the 17 items making up the SIGH-D-17. Each item is scored on a 3, 4, or 5-point scale. The maximum possible total score is 53. If any one of the 17 items is not scored (ie, has a

missing value), the total score will be set equal to missing. Note that a score of 3 for Item 8 (loss of weight) represents "not assessed", and should be ignored in calculating the total score.

The total score at each visit (screening, Day -1, and Weeks 2, 4, 6, 8, and 10) will be summarized with descriptive statistics by treatment group. Changes from baseline (Day -1) at each postbaseline visit will also be summarized.

#### 3.16.10. Prior and Concomitant Medications

Prior medications and concomitant medications will be summarized by WHO Drug Anatomical Therapeutic Chemical Classification (ATC) Level 3 category (or Level 2 if there is not an applicable Level 3 category) and preferred name.

Medications will be assigned to one or two study periods (prestudy or during screening vs. during the treatment period or posttreatment, follow-up period) based on the medication start and stop dates relative to the study drug dosing. For example, medications that were started and stopped prior to the date of the first dose of study drug will be assigned to the prestudy/screening period only, while medications started prior to the first dose of study drug and either stopped during the study or indicated as "ongoing" will be assigned to both the prestudy/screening and treatment/follow-up periods. A given medication can therefore be assigned to one or two study periods in the tabular summaries, depending on its start and end dates.

The number and percentage of subjects using medications in each WHO Drug ATC category (Level 3/preferred name) will be summarized by treatment group and study period as described in the next paragraph. A subject may take the same medication more than once or multiple medications for a subject may be classified under the same ATC level or preferred name. A subject is counted only once for each level of medication classification within a summary.

The summary of medications taken prestudy or during screening will be presented by treatment group. An "all subjects" column will be included in this summary. Medications taken during the study after the initiation of dosing (ie, during the treatment or follow-up periods) will be summarized by treatment group.

#### 3.17. Additional Data Presentations

#### 3.17.1. Inclusion and Exclusion Criteria

Inclusion and exclusion criteria confirmation results will be presented in a data listing by subject.

#### 3.17.2. Serology Test Results

Serology assessments (ie, Human immunodeficiency virus antibody [HIV-Ab], Hepatitis B surface antigen [HBsAg], and Hepatitis C antibody [HCV-Ab]) collected at screening will be reviewed at the study site to ensure the entry criteria are met. The HBsAg and HCV-Ab test results will be presented in a listing by subject. The results of the HIV-Ab test will not be listed, but will be kept on file at the study site.

# 3.17.3. Pregnancy Test Results

Serum and urine pregnancy test results will be presented in a listing by subject.

# 3.17.4. Urine Drug Screen and Alcohol Breath Test

Urine drug screen and alcohol breath test results will be presented in a listing by subject.

### 4. DEVIATIONS FROM PROTOCOL PLANNED ANALYSIS

The methods of analysis described in this SAP are generally consistent with the statistical methods described in the clinical study protocol (Amendment 3). The methods of analysis have been changed for two efficacy endpoints: the CGI-TS-Improvement score and the RTRS total score. The MMRM analysis was specified in the protocol for both of these endpoints. In this SAP, the ANOVA is specified for the CGI-TS-Improvement score, and the ANCOVA is specified for the RTRS total score. Sensitivity analyses have been added to the SAP for the primary efficacy endpoint. In addition, the CGI-TS-Improvement score mean change from baseline to Week 8 has been identified as the key secondary efficacy endpoint, and the fixed-sequence testing procedure has been included. The SAP includes additional endpoints and data summaries not mentioned in the study protocol, including the TTS responder analysis and the PCS value summaries for clinical laboratory data and vital signs.

# 5. PERFORMANCE QUALIFICATION OF SAS® PROGRAMS

The analysis and summary of data from this study will be performed using SAS® 9.3 (or a later release if available). All SAS® programs used in the production of statistical analyses, tables, listings, and figures described in this SAP will undergo performance qualification (verification that the program produces the intended output) in accordance with department standard operating procedures. The performance qualification may include independent programming and/or peer review of the SAS® log files. In addition, tables, figures, listings, and statistical analysis output will be independently reviewed for completeness and accuracy.

### 6. REFERENCES

ClinicalTrials.gov Identifier: NCT01727700. Otsuka Pharmaceutical Development & Commercialization, Inc. Study evaluating the safety and efficacy of fixed-dose once-daily aripiprazole in children and adolescents with Tourette's Disorder <a href="https://www.clinicaltrials.gov/ct2/show/NCT01727700?term=NCT01727700&rank=1">https://www.clinicaltrials.gov/ct2/show/NCT01727700?term=NCT01727700&rank=1</a> [Accessed 05 June 2015].

Jankovic J, Jimenez-Shahed J, Brown LW. A randomised, double-blind, placebo-controlled study of topiramate in the treatment of Tourette syndrome. J Neurol Neurosurg Psychiatry. 2010 Jan;81(1):70-3.

LaVange LM. The role of statistics in regulatory decision making. Therapeutic Innovation and Regulatory Science. 2014; 48(1) 10-19.

O'Kelly M, Ratitch B. Clinical Trials with Missing Data: A Guide for Practitioners. West Sussex, United Kingdom: John Wiley & Sons, Ltd. 2014; 292-297, 309-310.

Yoo HK, Joung YS, Lee JS, Song DH, Lee YS, Kim JW, et al. A multicenter, randomized, double-blind, placebo-controlled study of aripiprazole in children and adolescents with Tourette's disorder. J Clin Psychiatry. 2013;74(8):e772-80.